CLINICAL TRIAL: NCT05238298
Title: Efficacy and Mechanism of Repeated Transcranial Magnetic Stimulation in Children With Autism Spectrum Disorder: an Open-label Clinical Trial
Brief Title: Efficacy and Mechanism of rTMS in Children With ASD: an Open-label Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Fei Li, Chief Physician ,Doctoral Supervisor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2022-008
Record Dates: First submitted 2022-01-29; First posted 2022-02-14 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Repetitive Transcranial Magnetic Stimulation（rTMS）; Continuous theta Burst Stimulation （cTBS）
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rTMS Group (Experimental): Participants will receive continuous theta burst stimulation (cTBS) for a 10-day period (10 sessions). If feasible for the participant, all stimulation sessions will be held at the same time of the day.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — A technique that involves the use of electrical coils on the head to generate a brief magnetic field which reaches the cerebral cortex.

SUMMARY:
This study is a 6-week open-label clinical trial involving 20 children aged 6-10 years with autism spectrum disorder. During the study, subjects received repeated transcranial magnetic stimulation（rTMS）intervention at the left primary motor cortex (M1) 5 times per day for 10 days. From the beginning of intervention to the end of 4 weeks after the completion of intervention, the subjects's clinical symptomatology, cognitive psychology, neuroimaging, and adverse events will be followed up.Our purpose is to explore whether rTMS can improve the clinical symptoms of children with autism spectrum disorder in China, and to explore the neurophysiological mechanism of rTMS for autistic children.

DETAILED DESCRIPTION:
Participants will receive continuous theta burst stimulation (cTBS) for a 10-day period (10 sessions). If feasible for the participant, all stimulation sessions will be held at the same time of the day. During this study，participants' clinical symptomatology, cognitive psychology, neuroimaging, and adverse events will be followed up for four times, specifically，before intervention, 5 days after intervention, immediately after the completion of intervention , and 4 weeks after the completion of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-10 years.
* Meeting the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders, Edition 5 (DSM-5) .
* Confirmed by the ADOS and/or ADI-R diagnostic tool.
* IQ ≥70.
* Informed consent.

Exclusion Criteria:

* Patients with metal implants .
* Patients with neurological diseases such as epilepsy .
* Patients requiring surgical treatment due to structural abnormalities indicated by brain MRI .
* Genetic or chromosomal abnormalities .
* Suffering from mental disorders (such as mood disorders, etc.)
* Suffering from serious heart disease .
* Hearing-impaired .
* Intracranial hypertension .
* Participating in other clinical trials.
* Participants who received other interventions within 4 weeks prior to enrollment.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Social Response Scale (SRS) | Before intervention, 5 days after intervention, immediately after the completion of intervention , and 4 weeks after the completion of intervention
  SRS is a questionnaire used to assess the presence and severity of social impairment, with high scores indicating severe symptoms. Change of the SRS from baseline to 3 month after treatment to evaluate the effect of computer social interaction treatment on ASD children.

SECONDARY OUTCOMES:
Repetitive Stereotyped Behavior - Revised (RBS-R) | Before intervention, 5 days after intervention, immediately after the completion of intervention , and 4 weeks after the completion of intervention
  The Repetitive Behaviors Scale - Revised (RBS-R) is a 44-item self-report questionnaire that is used to measure the breadth of repetitive behavior in children, adolescents, and adults with Autism Spectrum disorders. The RBS-R provides a quantitative, continuous measure of the full spectrum of repetitive behaviors. The RBS-R consists of six subscales including: Stereotyped Behavior, Self-injurious Behavior, Compulsive Behavior, Routine Behavior, Sameness Behavior, and Restricted Behavior, that have no overlap of item content.
ADHD Rating Scale | Before intervention, 5 days after intervention, immediately after the completion of intervention , and 4 weeks after the completion of intervention
  ADHD Rating Scale is the most widely used ADHD screening and treatment monitoring tools.
Behavior Rating Inventory of Executive Function(BRIEF) | Before intervention, 5 days after intervention, immediately after the completion of intervention , and 4 weeks after the completion of intervention
  Specifically the investigators will evaluate the changes in executive function (EF) scores before and after cTBS treatment. The higer scores indicate more impairment in executive function.
Childhood Autism Rating Scale (CARS) | Before intervention, immediately after the completion of intervention , and 4 weeks after the completion of intervention
  CARS is a behaviour-rating scale used to assess the presence and severity of the symptoms of autism spectrum disorder(ASD), with scores ranging from 15 to 60 and high scores indicating severe symptoms. Change of the CARS from baseline to 3 months after treatment to evaluate the effect of tablet computer social interaction treatment on ASD children.
Clinical Efficacy Rating Scale (CGI) | 5 days after intervention, immediately after the completion of intervention , and 4 weeks after the completion of intervention
  CGI is a scale used to assess the severity of the illness and the global improvement of the patient under intervention.

OTHER OUTCOMES:
Cambridge Neuropsychological Test Automated Battery (CANTAB) | Before intervention, 5 days after intervention, immediately after the completion of intervention , and 4 weeks after the completion of intervention
  CANTAB tests have demonstrated sensitivity to detecting changes in neuropsychological performance and include tests of working memory, learning and executive function; visual, verbal and episodic memory; attention, information processing and reaction time; social and emotion recognition, decision making and response control.
Continuous Operation Test (CPT) | Before intervention, 5 days after intervention, immediately after the completion of intervention , and 4 weeks after the completion of intervention
  To obtain reliable parameters of behavior, continuous performance tasks (CPTs) are usually used where the subject performs a constant-difficulty task for minutes or tens of minutes without interruptions.
Resting State Electroencephalography | Before intervention, 5 days after intervention, immediately after the completion of intervention , and 4 weeks after the completion of intervention
  There are three main parameters: phase locking value(PLV) , coherence (Coh) and the power spectral density of alpha band (PSD). PLV and Coh are estimated for exploring the functional connectivity between the targeted brain region and the rest regions of brain.
Functional Near Infrared Spectroscopy , fNIRS | Before intervention, 5 days after intervention, immediately after the completion of intervention , and 4 weeks after the completion of intervention
  Head fNIRs is a non-invasive, non-ionizing method for measuring and imaging the functional hemodynamic response to brain activity. It measures changes in hemoglobin (Hb) concentrations within the brain by means of the characteristic absorption spectra of Hb in the near-infrared range. Changes in the head fNIRs results of the subject before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, Director, Principal Investigator — Xinhua hospital Affilated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- ShanghaiXinhua, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No